CLINICAL TRIAL: NCT04491162
Title: The Effect of Body Weight Support Treadmill Training on Lower Limb Function in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INK/ Rehab/ BWS/2016
Record Dates: First submitted 2020-05-18; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Gait Disorder, Sensorimotor
Keywords: Rehabilitation; Body weight supported treadmill training
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The observer was not allowed to know the treatment allocation. The patients were instructed not to discuss anything regarding his/ her treatment allocation with the examining investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional gait therapy (Active Comparator): Conventional gait therapy.
  Interventions: Other: Conventional therapy
- BWST training (Experimental): Conventional gait therapy + Body weight support treadmill training
  Interventions: Other: Body weight support treadmill training + conventional therapy

INTERVENTIONS:
Other: Body weight support treadmill training + conventional therapy — Conventional gait therapy was done based on the principles of the proprioceptive neuromuscular facilitation (PNF) and Motor Relearning program (MRP) concepts.
  Patients in intervention arm were additionally trained with a 40% body weight support and a comfortable walking speed on treadmill for twenty minutes. The training, which was conducted three times a week, for period of two weeks.
  Arms: BWST training
Other: Conventional therapy — Conventional gait therapy was done based on the principles of the proprioceptive neuromuscular facilitation (PNF) and Motor Relearning program (MRP) concepts.
  Arms: Conventional gait therapy

SUMMARY:
Stroke has severe debilitating neurological consequences for the victim. Within context of this study, gait disturbance is induced by disabilities in muscle weakness, abnormal muscle contraction, or postural control. Gait disturbance has an unfavorable effect on functional independence and prognosis of patients. Due to this reason, recovery in gait ability of stroke patients is considered as a very important goal in rehabilitation.

Body weight supported treadmill training (BWSTT) is a task-oriented technique for gait restoration after stroke. The present study focused on the possibility of BWSTT as a special program for improving gait ability. The purpose of this study was to evaluate the effectiveness of a BWSTT intervention useful as a short-term intensive program for chronic stroke survivors.

DETAILED DESCRIPTION:
Stroke is thought to be a serious health problem which can cause severe disabilities. Aspects of disabilities caused by stroke are various according to the affected region and its severity. In general, sensory deficits, cognitive problem, motor impairment, visual perceptual disorders and dysphagia mainly occur among stroke patients. In particular, gait disturbance is induced by disabilities in muscle weakness, abnormal muscle contraction, or postural control. This gait disturbance is exhibited as an asymmetric gait pattern, such as a decrease in paretic side stance phase and non-paretic swing phase, cadence, velocity and difference in step length and stride length. Therefore, these differences create abnormal gait patterns in stroke patients. Furthermore, gait disturbance has an unfavorable effect on functional independence and prognosis of patients. Due to this reason, recovery in gait ability of stroke patients is considered as a very important goal in rehabilitation.

Gait performance is an indicator of mobility impairment and disability after stroke. It predicts mortality, morbidity, and risk of future stroke. Gait speed is responsive to short-term rehabilitation. An improvement in gait speed of 0.16 m/s can reduce the level of assistance in patients with subacute stroke and was recommended to be the minimum clinically significant difference. The control of gait involves the planning and execution from multiple cortical areas, such as secondary and premotor cortex. Stroke patients often have gait impairment such as decreased gait speed and asymmetrical gait cycle as a result of cortical reorganization. Repetitive mass motor task practice had been shown to facilitate neuroplasticity and brain reorganization in stroke patients, resulting in enhanced motor recovery after stroke.

Body weight supported treadmill training (BWSTT) is a task-oriented technique for gait restoration after stroke. BWSTT has the advantage over conventional therapy as it offers higher intensity, more repetitive and task-oriented practice over the same period of time when compared to conventional therapy. Several studies have showed that BWSTT was more effective in gait speed improvement than regular physiotherapy. It has been demonstrated that BWSTT induces changes in corticomotor excitability which lead to improved balance and gait performance with chronic stroke. However, other studies have reported that BWSTT was not superior to conventional gait training.

Recent studies have reported that BWSTT can increase walking endurance in the subacute stage after stroke, but no improvement was reported in balance and 10 m gait speed. To date, there are very few studies that have used gait analysis to show how the improvements in gait parameters come about after BWSTT or conventional therapy. There is still a lack of basic understanding of gait training on human locomotion.

Despite substantial recovery of independent ambulation by survivors following unilateral stroke, persistent gait abnormalities are observed in a large percentage of these persons. In these circumstances, a short-term intermittent and intensive rehabilitation program for chronic stroke survivors is thought to be particularly efficient for shoring up their independence, and the present study focused on the possibility of BWSTT as a special program for improving gait ability. The purpose of this study was to evaluate the effectiveness of a BWSTT intervention useful as a short-term intensive program for chronic stroke survivors.

ELIGIBILITY:
Inclusion criteria

* Age between 18 and 69 years, both genders will be acceptable.
* First episode of supratentorial stroke in hemiparesis (both ischaemic and haemorrhagic strokes)
* After 6 month from onset of stroke.
* All subjects were ambulatory before stroke
* Able to understand and follow simple verbal instruction, scoring at least 24 out of 30 on Mini Mental State Examination.
* Able to walk at least 10 meters distance independently, with or without a walking aids.
* Walking speed<0.75m/s at their self-selected velocity (SSV).
* Scoring 3 or 4 in Functional Ambulation Category Scale.
* Scoring less than 21 out of 23 on trunk Impairment Scale.
* Currently not receiving any other type of physiotherapeutic intervention.

Exclusion criteria

* Neurological disease affecting balance other than stroke.
* History of diagnosed musculoskeletal disorder of the trunk and / or lower extremities affecting the motor performance.
* History of Cerebrovascular accident more than one time or bilateral CVA at a time.
* Myocardial infarction within the past 6 months.
* Angina or ischemia at rest or during exercise.
* Unstable hypertension (>150/90 mmHg), arrhythmia, congestive heart failure or unstable cardio vascular status.
* Absence of active movement in the paretic lower limbs.
* Disability of joint including hip fracture and severe cardio pulmonary disease.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
10 meter walk test | Two weeks
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.

SECONDARY OUTCOMES:
Cadence | Two weeks
  Cadence is measured as number of steps per minute during a 10 metre walk.
Timed up and go test | Two weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Berg Balance Scale | Two weeks
  It is a widely used clinical test for static and dynamic balance. It comprises of 14 balance related tasks. A score of less than 20 signifies wheelchair use; 20-40: walking with assistance; 40-56: Independent ambulator.

CONTACTS AND LOCATIONS:
Overall Officials: Madhusree Sengupta, MD, PDF, Principal Investigator — Consultant
Locations (1):
- Institute of Neurosciences Kolkata, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No